CLINICAL TRIAL: NCT01247246
Title: A Phase 2b, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Three Different Doses of SCV 07 in Attenuating Oral Mucositis in Subjects With Head and Neck Cancer Receiving Concurrent Chemotherapy and Radiotherapy
Brief Title: Study to Evaluate the Efficacy and Safety of Three Different Doses of SCV 07 in Attenuating Oral Mucositis in Subjects With Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCI-SCV-MUC-P2b-002
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Oral Mucositis
Keywords: Oral Mucositis; Head and Neck; Head and Neck Neoplasms; Mucositis; Stomatitis; Neoplasms by Site; Neoplasms; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Mouth Diseases; Stomatognathic Diseases; SCV-07
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Mucositis; Neoplasms by Site; Neoplasms; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Mouth Diseases; Stomatognathic Diseases | interventions — golotimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- SCV-07 0.1mg/kg (Active Comparator)
  Interventions: Drug: SCV-07
- SCV-07 0.3mg/kg (Active Comparator)
  Interventions: Drug: SCV-07
- SCV-07 1.0mg/kg (Active Comparator)
  Interventions: Drug: SCV-07

INTERVENTIONS:
Drug: SCV-07 — clinical trial material; (placebo or SCV 07) at doses of 0 (placebo), 0.1, 0.3, and 1.0 mg/kg will be administered sc
  Arms: SCV-07 0.1mg/kg; SCV-07 0.3mg/kg; SCV-07 1.0mg/kg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a phase 2b, double-blind, placebo-controlled, 4-arm, adaptive-design trial, initially stratified by cisplatin regimen, and then randomized 1:1:1:1. The study will be conducted in subjects receiving ChemoRT for the treatment of squamous cell carcinomas (SCCs) of the oral cavity, oropharynx, hypopharynx, or larynx. The study includes a treatment period of approximately 7 weeks, depending on the subject's prescribed radiation plan, and Week 1 and Week 4 post RT follow-up visits. It also includes a longer follow-up period of approximately 12 months to determine if there is an effect of SCV 07 on the tumor response to ChemoRT.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign an informed consent form (ICF) for the study approved by the Investigator's local or a central Institutional Review Board (IRB)
* Have recently diagnosed, pathologically confirmed, non-metastatic SCC of the oral cavity, oropharynx, hypopharynx, or larynx that will be treated with ChemoRT as first-line treatment; subjects with a history of surgical management are eligible
* Have a plan to receive a continuous course of conventional external beam irradiation delivered by intensity-modulated radiotherapy (IMRT) as single daily fractions of 2.0 to 2.2 Gy, with a cumulative radiation dose between 50 and 72 Gy. Planned radiation treatment fields must include at least 2 oral sites (buccal mucosa, floor of oral cavity, tongue, or soft palate), with each site receiving ≥ 50 Gy
* Have a plan to receive a standard cisplatin CT regimen administered tri-weekly (80 to 100 mg/m2, on Days 0, 21, and 42) or weekly (30 to 40 mg/m2)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Have adequate hematopoietic, hepatic, and renal function at the screening visit:

  * Hematopoietic function

    * Hemoglobin ≥ 10 g/dL
    * Absolute neutrophil counts (ANC) ≥ 1,500 cells/mm3
    * Platelet count ≥ 100 × 109/L
  * Hepatic function

    * Total bilirubin < 1.5 times the upper-normal limit (ULN)
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 times the ULN
  * Renal function: Serum creatinine concentration ≤ 2 mg/dL; if result is ≥ 1.4 mg/dL and ≤ 2.0 mg/dL, a 24-hour urinary creatinine clearance test must be performed by the site's local laboratory. To be eligible for the study, a subject must demonstrate a 24-hour urinary creatinine clearance ≥ 50 mL/min
* Have a negative serum pregnancy test if a woman is of childbearing potential
* Agree to use medically acceptable methods of birth control during study participation and for 30 days following the last CTM treatment if a woman is of childbearing potential
* Males or females aged 18 years or older.

Exclusion Criteria:

* Tumor of the lips, sinuses, salivary glands, nasopharynx, or unknown primary tumor
* Metastatic disease (M1) Stage IV C
* Prior radiation to the head and neck
* Plan to be treated with cetuximab (Erbitux®)
* Have undergone induction CT
* History of other malignant tumors, excluding non-melanoma skin cancer or curatively excised in situ cervical carcinoma
* Have had a major surgical procedure, other than for HNC, or significant traumatic injury within 4 weeks prior to the initiation of RT; anticipation of need for a major surgical procedure during the study
* Active infectious disease, excluding oral candidiasis
* Have OM at the baseline visit
* Have a diagnosis of autoimmune disease requiring chronic immunosuppression
* Known seropositivity for HIV, HBV, or HCV
* Prior use of SCV 07
* Have used any investigational agent within 30 days of randomization
* Are pregnant or breastfeeding
* Known allergies or intolerance to cisplatin
* Unable to give informed consent or comply with study requirements, including completing the subject diary and QOL instruments
* Have any other condition or therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy | June 2012
  The primary objective of the study is to evaluate the efficacy of SCV 07 in modifying the course of oral mucositis (OM) in subjects with head and neck cancer (HNC) receiving concurrent ChemoRT.

SECONDARY OUTCOMES:
Safety | June 2012
  The secondary objective of the study is to evaluate the safety and tolerability of SCV 07.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Rios, MD, Study Director — SciClone Pharmaceuticals
Locations (49):
- United States (49):
  - Arizona Center for Cancer Care, Peoria, Arizona
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Disney Family Cancer Center, Burbank, California
  - City of Hope National Medical Center, Duarte, California
  - VA Long Beach Health System, Long Beach, California
  - Pomona Valley Hospital, Pomona, California
  - Yale University School of Medicine, New Haven, Connecticut
  - The Whittingham Cancer Center, Norwalk Hospital, Norwalk, Connecticut
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Lake County Oncology and Hematology, Tavares, Florida
  - The University of Illinois at Chicago, Chicago, Illinois
  - St. John's Cancer Center, Anderson, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital, Baltimore, Maryland
  - Southcoast Hospital Group, Fairhaven, Massachusetts
  - Gershenson Radiation, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - The Nebraska Medical Center, Omaha, Nebraska
  - Veterans Administration NJ Health Care System, East Orange, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Rochester University Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Memorial Hospital of Rhode Island Cancer Center, Pawtucket, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Cookeville Regional Cancer Center, Cookeville, Tennessee
  - Kirkland Cancer Center/Jackson Madison County General Hospital, Jackson, Tennessee
  - Tyler Hematology Oncology, Tyler, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Wheeling Hospital, Wheeling, West Virginia
  - Medical College of Wisconson, Milwaukee, Wisconsin

REFERENCES:
- See also: SciClone Pharmaceuticals, Inc. — http://www.sciclone.com